CLINICAL TRIAL: NCT03495895
Title: The Effectiveness of MInding the Baby in a Danish Community Sample
Acronym: MTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: Yale University (Other); Metodecentret - Center for Effective Innovation in Social Services (Unknown)
Responsible Party: Principal Investigator, Maiken Pontoppidan, Researcher, VIVE - The Danish Center for Social Science Research
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: VIVE
Record Dates: First submitted 2018-01-30; First posted 2018-04-12 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Family; Pregnancy, High Risk
Keywords: Disadvantaged families; Pregnancy; Intervention; Minding the Baby

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As the intervention is a home visiting intervention participants and care providers cannot be blinded. Outcome assessor and data analyst will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minding the Baby (Experimental): Families are visited weekly beginning in the mother's third trimester of pregnancy up through the child's first birthday, at which point visits take place biweekly up through the child's second birthday.
  Interventions: Behavioral: Minding the Baby
- Control (Other): Usual care control condition. Families in the control Group receive the usual care that is offered to families in the target group
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Minding the Baby — Visits are carried out on an alternating basis by a team made up of a nurse practitioner (NP) and social worker.
  Arms: Minding the Baby
Behavioral: Usual Care — Usual care condition
  Arms: Control

SUMMARY:
Minding the Baby is an intensive and preventive home-visiting programme that helps vulnerable or high risk mothers. MTB is delivered by an interdisciplinary team. Ten Danish sites will be randomized to training at time 1 or 2 and recruit usual care control families before they receive the training. Families are assessed before they give birth and when their child is three months, one and two years old with a range of assessments including maternal sensitivity, parent mental Health, child development, and health related register data. The aim of the trial is to assess the effectiveness of Minding the Baby to improve mother-child relations and the mental health of parents and children.

DETAILED DESCRIPTION:
Minding the Baby is an intensive and preventive home-visiting programme that helps vulnerable or high risk mothers. The focus of the intervention is to reduce negative infant and maternal outcomes and strengthen the attachment relationship. MTB is delivered by an interdisciplinary team of highly skilled practitioners, who have health and social work experience, integrating advanced practice nursing and mental health care for mothers and infants. In the proposed Randomised Control Trial (RCT) the investigators will study the efficacy of this innovative intervention across ten Danish sites. Site staff will be trained at two sessions one year apart. Sites are randomized to training at time 1 or 2. All sites will recruit treatment as usual control families before they receive the training and start offering the intervention to all families. Potential participants will be approached by a local front staff member (e.g. midwife, helath visitor or social worker) who will inform mothers of the project in the early pregnancy. Consenting eligible participants will be assessed before they give birth and when their child is three months, one and two years old.

The effectiveness of the MTB programme will be evaluated by assessing a range of maternal and infant outcomes, including maternal sensitivity, parent mental Health, child development, and register data on e.g. infant maltreatment and neglect, hospitalization, income, immunization. By combining parent report, observational and register data researchers will get a unique opportunity to advance knowledge regarding effective ways to support some of the youngest and most vulnerable children in Denmark.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant vulnerable women

Exclusion Criteria:

* Current severe substance abuse
* Severe psychotic illness
* Profound or severe learning disabilities
* Life-threatening illness in parent or child
* Non-Danish speaking

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Maternal sensitivity measured by the CIB (Coding Interactive Behavior) | at child age 24 months
  Maternal sensitivity

SECONDARY OUTCOMES:
Maternal sensitivity measured by the CIB (Coding Interactive Behavior) | Child age 12 months
  Maternal sensitivity
Coding interactive bahavior (CIB) | child age 12 and 24 months
  Parent child relationship Subscales: Intrusiveness, Limit setting, Involvement, Withdrawal, Reciprocity, Negative states
Ages and Stages Questionnaire-Social Emotional 2 (ASQ:SE-2) | 3, 12 and 24 months
  Child social-emotional Development Total score range 0-150 ( 3 months 15 items), 0-260 (12 months 26 items), 0-300 (24 months 30 items). Low score is better.
Edinburgh Postnatal depression Scale (EPDS) | 3, 12 , 24 months
  Depression Total score range 0-30. Low score is better
Warwick-Edinburgh Mental Well-being Scale | Baseline, 3, 12 , 24 months
  Maternal mental Health 7 items. A total score i calculated by summing the 7 items and converting the raw score according to a published conversion table. Raw score range 7- 35. Converted score range 7-35. High is better outcome.
2-5 | 24 months
  The name of the measure is 2-5 and measures child Development. Subscales included: Perception (7 items) low score is better, Language (10 items) low score is better
Prenatal Parental reflective functioning questionnaire (P-PRFQ) | Baseline
  Parental reflective functioning for pregnant women. Total score range 14-98. Higher score is better. Three subscales: Opacity of mental states (4 items), reflecting on the fetus-baby (3 items) and Dynamic of mental states (5 items)
Parental reflective functioning questionnaire (PRFQ-1) | 12 and 24 months
  Parental reflective functioning Three subscales score range 6-42: Pre-Mentalizing Modes (PRFQ-PM) 6 items. low score is better. Certainty about Mental States (PRFQ-CMS) 6 items high score is better. Interest and curiosity in mental states PRFQ-IC 6 items high score is better.
Parental Stress Scale (PSS) | 12 ,24 months
  Parental stress Total score range 18-90 low score is better
Ages and Stages Questionnaire 3 (ASQ:3) | 3 months
  Child development
Acitvities with child | 12 and 24 months
  Singing and reading Total score range 0-70. High score is better.
SEAM Family profile | 12 months
  Family profile
Parent behavior Inventory (PBI) | 12 and 24 months
  Parent Behavior. Two subscales Supportive/Engaged and Hostile/Coercive.
Being a Mother (BAM-13) | 3 months
  Maternal confidence. Total score range 0-39. Low score is better
Hospital Anxiety and Depression Scale (HADS) | Baseline, 3, 12,24 months
  Two subscales Anxiety (range 0-21 low score is better) and depression (range 0-21 low score is better)
PTSD-8 | Baseline, 12 and 24 months
  A Short PTSD Inventory. Total score range 8-32, low score is better
Experiences in Close Relationship Scale-Short Form (ECR-S) | Baseline, 12, 24 months
  Two subscales Anxiety (range 1-42 low score is better) and Avoidance (range 1-42 low score is better)

CONTACTS AND LOCATIONS:
Overall Officials: Maiken Pontoppidan, Ph.D., Principal Investigator — VIVE
Locations (1):
- VIVE - The Danish Centre of Applied Social Science, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
There will be few participants from each local authority and data can therefore not be made publicly available due to protect participant privacy

REFERENCES:
- [Derived] Pontoppidan M, Hirani JC, Friis-Hansen M. Minding the Baby versus usual care: effects on parental sensitivity and parent-child interaction in a cluster quasi-randomized trial. Attach Hum Dev. 2025 Aug;27(4):567-590. doi: 10.1080/14616734.2025.2534608. Epub 2025 Jul 28. PMID 40717494
- [Derived] Pontoppidan M, Thorsager M, Friis-Hansen M, Slade A, Sadler LS. Minding the Baby versus usual care: study protocol for a quasi-cluster-randomized controlled study in Denmark of an early interdisciplinary home-visiting intervention for families at increased risk for adversity. Trials. 2022 Jun 24;23(1):529. doi: 10.1186/s13063-022-06434-2. PMID 35751089